CLINICAL TRIAL: NCT00061126
Title: A Clinical Trial Evaluating the Safety and Efficacy of ABX-EGF in Patients With Hormone Resistant Prostate Cancer With or Without Metastasis
Brief Title: ABX-EGF (a Monoclonal Antibody) Given to Patients With Prostate Cancer With or Without Tumor in Other Parts of the Body
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abgenix (Industry)
Collaborators: Immunex Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX-0310; ABX-EGF
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PSA; Hormone refractory; Rising PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Panitumumab

INTERVENTIONS:
Drug: ABX-EGF

SUMMARY:
A clinical trial examining the safety and effectiveness of ABX-EGF when given to patients with prostate cancer with or without tumor in other parts of the body.

Patients will be treated for a maximum of 48 doses (6 treatment courses; 8 doses per course) or until evidence of progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years of age or older
* Has tumor tissue available for diagnostics
* Failed front line luteinizing hormone-releasing hormone analogue (LHRH) such as leuprolide or goserelin, or failed orchiectomy, as evidenced by disease progression. Patients must continue on a LHRH analogue (unless the patient had an orchiectomy) throughout the course of the study
* ECOG score of 0 or 1

Exclusion Criteria:

* Any prior chemotherapy for prostate cancer besides hormonal therapy (including no prior EGFr targeting agent)
* Prior history of cancer other than prostate carcinoma within the past 5 years that has required treatment or been active (prior basal cell carcinoma is allowed)
* Known to be HIV positive
* Myocardial infarction within one year prior to entering the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA School of Medicine, Los Angeles, California
  - Stanford Medical Center, Stanford, California
  - Advanced Research Institute, New Port Richey, Florida
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Urology San Antonio Research, San Antonio, Texas
  - University of Washington, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington